CLINICAL TRIAL: NCT07177911
Title: A Phase I Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Immunogenicity of CC312 in Patients With Moderate-to-Severe Systemic Lupus Erythematosus
Brief Title: Safety and Efficacy Study of CC312 for Moderate to Severe SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CytoCares Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC312-S-001
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: SLE - Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CC312 (Experimental)
  Interventions: Drug: CC312
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC312 — Subjects will initially receive a single intravenous dose of CC312. After a 21-day period following the first dose, the patient may proceed to the multiple intravenous dosing phase only after investigators and the sponsor have confirmed acceptable safety and tolerability.
  Arms: CC312
Drug: Placebo — Subjects will initially receive a single intravenous dose of Placebo. After a 21-day period following the first dose, the patient may proceed to the multiple intravenous dosing phase only after investigators and the sponsor have confirmed acceptable safety and tolerability.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled Phase I clinical trial featuring single and multiple ascending doses. It is designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, and preliminary efficacy of CC312 in adult patients with moderate to severe systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the trial's purpose, nature, methodology, and potential adverse reactions, voluntarily participate as a subject, and sign the informed consent form.
* Aged 18 to 65 years (inclusive, based on the date of signing the informed consent form), regardless of gender.
* Diagnosed with systemic lupus erythematosus (SLE) according to the 2019 EULAR/ACR classification criteria.
* SLEDAI-2000 score ≥7 with at least one BILAG A or two BILAG B domains, despite standard therapy.
* Meet at least one of the following criteria: positive antinuclear antibody (ANA) ≥1:80 at screening, positive anti-dsDNA antibody at screening, or positive anti-Sm antibody at screening.
* Have had an inadequate response to at least two standard therapies (e.g., corticosteroids, antimalarials, immunosuppressants, biologics) prior to screening, including at least one immunosuppressant and/or biologic. Prior to the first dose, subjects must have been on a stable dose of corticosteroids (e.g., ≤40 mg/day prednisone or equivalent at screening and during the screening period; if used alone, ≥7.5 mg/day prednisone or equivalent) and/or antimalarials and/or immunosuppressants for at least 12 weeks, with doses stable for ≥30 days.
* Females of childbearing potential must agree to use highly effective contraception from screening until 6 months after the last dose and refrain from oocyte collection or donation during this period. Their male partners of childbearing potential must also use effective contraception.
* Males of childbearing potential must agree to use highly effective contraception from screening until 6 months after the last dose, with no plans for fertility or sperm donation. Their female partners of childbearing potential must also use effective contraception during this period.

Exclusion Criteria:

* Severe lupus nephritis within 8 weeks prior to screening (defined as urinary protein >6 g/24 h, or serum creatinine >2.5 mg/dL or 221 μmol/L, or requiring prohibited medications for active nephritis per protocol, or needing hemodialysis, or receiving prednisone ≥100 mg/d or equivalent glucocorticoids for ≥14 days).
* Central nervous system disorders (including but not limited to epilepsy, psychosis, interstitial encephalopathy syndrome, cerebrovascular accident, encephalitis, CNS vasculitis) within 8 weeks prior to screening, whether SLE-related or not.
* History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
* Other concurrent autoimmune diseases requiring systemic therapy, except for Sjögren's syndrome.
* IgA deficiency (serum IgA level <10 mg/dL).
* Abnormal laboratory findings at screening:

Liver function: AST/ALT or total bilirubin >2× upper limit of normal (ULN); Hematology: hemoglobin <85 g/L, WBC <2.5×10⁹/L, neutrophil count <1.0×10⁹/L, platelet count <50×10⁹/L; Renal function: eGFR <30 mL/min/1.73 m²;

* Participation in any other clinical trial (including cell or gene therapy) within 4 weeks prior to screening or within 5 half-lives of the investigational product (whichever is longer).
* Received CAR-T therapy within 6 months prior to screening.
* Treatment with B-cell-depleting agents (e.g., rituximab, or therapies targeting CD19/CD20/BAFF) within 6 months prior to screening, unless B-cell levels have returned to pre-treatment or normal ranges.
* Received non-standard anti-SLE therapies (e.g., Saphnelo) within 3 months or 5 half-lives of the drug (whichever is longer) prior to screening.
* Received live/attenuated vaccination within 4 weeks prior to screening or plans to receive such during the trial.
* Active infection within 14 days prior to screening (bacterial, viral, fungal, parasitic, or other).
* History of Grade 3-4 allergic reaction (per CTCAE v5.0) to another monoclonal antibody, or known hypersensitivity to any component of CC312 (including recombinant proteins, polysorbate 80, etc.). Patients with transient (≤24 h) Grade ≤3 reactions may be included after discussion with the investigator.
* Evidence of drug abuse, substance abuse, or alcohol addiction.
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to screening; wounds must be fully healed (procedures like catheter placement are excluded).
* History of cardiovascular events within 6 months prior to screening: NYHA Class III/IV heart failure, myocardial infarction, unstable angina, uncontrolled/symptomatic atrial arrhythmia, ventricular arrhythmia, or other clinically significant cardiac conditions.
* Any other severe underlying disease (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular events, GI bleeding, severe coagulation disorders), psychiatric disorder, or social circumstances that may interfere with trial conduct, compliance, or pose high risk per investigator's judgment.
* Concurrent malignancy diagnosed within <5 years prior to screening.
* Grade ≥2 bleeding within 30 days prior to screening, or requiring long-term anticoagulants (e.g., warfarin, LMWH, factor Xa inhibitors).
* Pregnant or lactating women.
* Positive screening for: tuberculosis (PPD skin test or TB-IGRA, unless with prior adequate anti-TB treatment and no current signs), HIV antibody, HBsAg or HBcAb, HCV antibody, or TP antibody.
* Any other condition deemed ineligible by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-11 (Estimated); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE)/serious adverse events (SAE) | 2 years
  All adverse events will be evaluated and graded according to the severity criteria of CTCAE (Common Terminology Criteria for Adverse Events) version 5.0, with the exception of Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS), which will be assessed using the ASTCT (American Society for Transplantation and Cellular Therapy) standard.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of CC312 | 2 years
  Blood samples will be collected for serum concentration analysis at specific time points
Area Under the Concentration-time Curve (AUC) of CC312 | 2 years
  The area under the concentration-time curve (AUC) was calculated using the linear trapezoidal rule.
Counts of peripheral B cells | 2 years
  Blood samples will be collected for CD19+ and CD20+ B cell subsets analysis at specific time points
Anti-double-stranded DNA antibody （anti-dsDNA antibody） | 2 years
  Blood samples will be collected at specific timepoints for anti-double-stranded DNA antibodies (anti-dsDNA) analysis.
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2000) score | 2 years
  SLEDAI-2000 score is used to evaluate the clinical symptoms and disease activity of SLE. The score ranges from 0 to 15, with higher scores indicating more severe disease activity.
Anti-CC312 Antibodies | 2 years
  Blood samples will be collected at specific time points to assess the immunogenicity of the drug, primarily through the detection of anti-CC312 antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murimi-Worstell IB, Lin DH, Kan H, Tierce J, Wang X, Nab H, Desta B, Alexander GC, Hammond ER. Healthcare Utilization and Costs of Systemic Lupus Erythematosus by Disease Severity in the United States. J Rheumatol. 2021 Mar;48(3):385-393. doi: 10.3899/jrheum.191187. Epub 2020 Jul 1. PMID 32611669
- [Background] Gergianaki I, Bortoluzzi A, Bertsias G. Update on the epidemiology, risk factors, and disease outcomes of systemic lupus erythematosus. Best Pract Res Clin Rheumatol. 2018 Apr;32(2):188-205. doi: 10.1016/j.berh.2018.09.004. Epub 2018 Sep 27. PMID 30527426
- [Background] Tsokos GC. Systemic lupus erythematosus. N Engl J Med. 2011 Dec 1;365(22):2110-21. doi: 10.1056/NEJMra1100359. No abstract available. PMID 22129255